CLINICAL TRIAL: NCT02363907
Title: Observational Study to Evaluate the Effectiveness and Safety of the Dexcom G4
Brief Title: Observational Study to Evaluate the Effectiveness and Safety of the Dexcom G4 Continuous Glucose Monitoring System in Pediatrics
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-900982
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2015-02

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; pediatric; continuous glucose monitoring system; CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the Dexcom G4 System when used as an adjuvant to blood glucose testing over a 7-day period in people 2 to 17 years-old with diabetes mellitus.

DETAILED DESCRIPTION:
Performance of the system will be primarily evaluated by comparing the blood glucose measurements from the reference device, a blood glucose meter, to the CGM System values collected during the study. Specifically, performance will be primarily evaluated in terms of the proportion of G4 System values that are within ±20% of glucose meter reference value for glucose levels >80 mg/dL and ±20 mg/dL of glucose meter reference values <80 mg/dL. These G4-meter matched pairs will be analyzed across the 7 days of wear.

Safety data of the CGM System will also be collected and safety will be characterized by the incidence of anticipated device-related adverse events (ADEs) of subjects who participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 17 years;
* Diagnosis of diabetes mellitus;
* Treatment of diabetes with insulin and/or oral diabetes medication Note: Insulin-using subjects only - willing to avoid insulin injections or wear an insulin pump insertion set within 3 inches from the sensor site;
* Willing to refrain from the use of medications containing acetaminophen during the sensor insertion period and for one day prior to sensor insertion;
* Able to perform up to 7 fingersticks per day during home use (approximately 2 calibration fingersticks or as often as prompted by the device and approximately 5 for diabetes management and/or detection of hyper and hypoglycemia); and
* Subject or guardian is able to speak, read, and write English.

Exclusion Criteria:

* Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
* Known allergy to medical-grade adhesives;
* For subjects of childbearing potential: are pregnant as demonstrated by a positive pregnancy test within 72 hours prior to device insertion;
* Hematocrit value outside the range of the blood glucose monitoring system used in the study;
* Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study);
* Planned MRI scan, CT scan, or diathermy during the week of the study; or
* Any condition that, in the opinion of the Investigator, would interfere with their participation in the trial (e.g., marked visual impairment) or pose an excessive risk to study staff handling venous blood samples (e.g., known history of hepatitis B or C, or HIV).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents with diabetes mellitus (Type 1 or Type 2)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Liljenquist, M.D., Principal Investigator — Rocky Mountain Diabetes and Osteoporosis Center
Locations (1):
- Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by one endocrinology practice in the US over a month long period, between Sep-Oct, 2012.
Groups:
- Single Arm- Performance, Using Blood Glucose Meter Reference: Subjects acting as their own control,comparing glucose values between CGM and blood glucose meters for %20/20 agreement
Period: Overall Study
Arm/Group | Single Arm- Performance, Using Blood Glucose Meter Reference
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Subjects acting as their own control,comparing glucose values between CGM and blood glucose meters for %20/20 agreement
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
Duration of diabetes [Mean (Standard Deviation); unit: years] | 4.3 (3.1)
Baseline A1C [Mean (Standard Deviation); unit: percent] | 8.6 (1.3)
CGM Experience Level [Mean (Standard Deviation); unit: years] | 0.2 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Point Accuracy of CGM ISF Readings to Blood Glucose Measured by a Reference Device
Description: "Point Accuracy was evaluated in terms of the percentage of CGM values that were within ±20% of glucose meter reference value for glucose levels >80 mg/dL and ±20 mg/dL of glucose meter reference values for glucose levels <80 mg/dL
Time Frame: Measured during clinic session during 7 day sensor wear period
Measure: Number (95% Confidence Interval); unit: Percentage of matched pairs w/i %20/20
Groups:
- Single Arm: Subjects as their own control, comparing ISF glucose readings to capillary blood glucose readings, measured by blood glucose meters
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Percentage of matched pairs w/i %20/20 | 77 [75 to 79]

ADVERSE EVENTS:
Groups:
- Single Arm,Performance, Using Blood Glucose Meter Reference: Subjects acting as their own control,comparing glucose values between CGM and blood glucose meters for %20/20 agreement
Arm/Group | Single Arm,Performance, Using Blood Glucose Meter Reference
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No